CLINICAL TRIAL: NCT05559671
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Non-inferiority Crossover Study Evaluating the Safety and Immunogenicity of the Herpes Zoster Subunit Vaccine in Patients With Systemic Lupus Erythematosus
Brief Title: Safety of the Herpes Zoster Subunit Vaccine in Lupus
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 22-00922
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Herpes Zoster Subunit Vaccine
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HZ/su Vaccine, then Placebo (Experimental): During the initial 24-week period (Period 1), participants will receive HZ/su injection at week 0 and week 8. During the second 24-week period (Period 2), participants will receive placebo saline injection at week 24 and week 32.
  Interventions: Biological: Herpes Zoster Subunit (HZ/su) Vaccine; Biological: Placebo
- Placebo, then HZ/su Vaccine (Experimental): During the initial 24-week period (Period 1), participants will receive placebo saline injection at week 0 and week 8. During the second 24-week period (Period 2), participants will receive HZ/su injection at week 24 and week 32.
  Interventions: Biological: Herpes Zoster Subunit (HZ/su) Vaccine; Biological: Placebo

INTERVENTIONS:
Biological: Herpes Zoster Subunit (HZ/su) Vaccine — Manufactured by GSK Biologicals SA. Administered as two-time injection of 0.5 mL each at either weeks 0 and 8 or weeks 24 and 32.
  Other Names: SHINGRIX
Biological: Placebo — Saline injection. Administered as two-time injection of 0.5 mL each at either weeks 0 and 8 or weeks 24 and 32.

SUMMARY:
This randomized, double-blind, placebo-controlled, non-inferiority crossover study will evaluate the Herpes Zoster Sunbit (HZ/su) vaccine in SLE patients in order to evaluate safety and immunogenicity in patients with variable baseline clinical activities, ages and immunosuppressant exposures. The investigators hypothesize that HZ/su administration will be non-inferior to placebo with respect to the risk of moderate or severe SLE flare(s) occurring within 24 weeks of receiving the first dose of the assigned treatment. In addition, the investigators hypothesize that immunogenicity of the vaccine in SLE patients will be at least 50% of levels observed in healthy subjects from prior large clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male ≥18 years of age at the time of signing the informed consent
3. Meet the 2019 EULAR/ACR Classification Criteria for SLE
4. Female subjects must use 1 effective method of avoiding pregnancy, from the time they sign consent until end of the study period unless the subject is surgically sterile (e.g., bilateral oophorectomy or complete hysterectomy), has a sterile male partner, is at least 1 year postmenopausal, or practices sustained abstinence consistent with the subject's customary lifestyle. Postmenopausal is defined as at least 1 year since last menses and the subject has an elevated follicle-stimulating hormone (FSH) level greater than the threshold laboratory value of post-menopausal women at screening.

Exclusion Criteria:

1. Prior administration of the Herpes Zoster subunit vaccine (Shingrix) or the Varicella-Zoster virus vaccine live (Zostavax)
2. Clinical HZ infection within 12 months prior to screening or during screening
3. Hybrid SLEDAI >12 at screening visit
4. Presence of a mild, moderate, or severe flare per the rSFI at time of screenin
5. Increase in clinical SLEDAI parameters at time of enrollment relative to screening visit
6. Any vaccine, including the final/booster dose of any SARS-CoV-2 vaccine, within six weeks enrollment
7. Receipt of rituximab or cyclophosphamide within nine months of enrollment
8. Participation in an interventional clinical trial of SLE or other therapeutics within six months of enrollment
9. Moderate to severe infectious febrile illness or use of systemic antibiotics (antibacterial, antiviral, antifungal, or antiparasitic agent) within 4 weeks of enrollment
10. Are pregnant, nursing, or planning a pregnancy while enrolled in the study
11. Known primary or secondary immunodeficiency (malignancy, HIV, common variable immune deficiency) or medications used during cancer chemotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of either Moderate or Severe Lupus Flares within 24 Weeks of First Dosing with HZ/su Vaccine | Up to Week 48
  Classification of moderate or severe lupus flares based on revised Safety of Estrogens in Lupus Erythematosus, National Assessment (SELENA) Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) Flare Index [rSFI].

SECONDARY OUTCOMES:
Occurrence of either Moderate or Severe Lupus Flares at Week 8 | Week 8
  Classification of moderate or severe lupus flares based on rSFI.
Occurrence of either Moderate or Severe Lupus Flares at Week 24 | Week 24
  Classification of moderate or severe lupus flares based on rSFI.
Occurrence of Mild, Moderate, or Severe Lupus Flares within 24 Weeks of First Dosing with HZ/su Vaccine | Up to Week 48
  Classification of mild, moderate, or severe lupus flares based on rSFI.
Occurrence of New or Worsening Disease Activity in Any Organ System as Identified by BILAG 2004 within 24 Weeks of First Dosing with HZ/su Vaccine | Up to Week 48
  The British Isles Lupus Assessment Group (BILAG) 2004 scores disease involvement within nine organ systems. Each of the 101 items are rated as 0 (not present), 1 (improving), 2 (same), 3 (worse), or 4 (new) in the last 4 weeks, compared with the previous 4 weeks.
Occurrence of Increase in PGA Score by More than 0.3 Points within 24 Weeks of First Dosing with HZ/su Vaccine | Up to Week 48
  Physician's Global Assessment (PGA) is a 10-cm visual analogue scale (VAS) anchored at 0 (none) and 3 (severe) with intermediate lines at 1 (mild) and 2 (moderate). Higher scores indicate greater severity of disease activity.
Occurrence of Grade 3 or Higher Adverse Events as Per CTCAE or Solicited AIT within 24 Weeks of First Dosing with HZ/su Vaccine | Up to Week 48
  Common terminology criteria for adverse events (CTCAE) and solicited assessments of intensity and toxicity (AIT) used to grade severity of adverse events.
Levels of Serum Varicella-Zoster Virus Anti-Glycoprotein E Antibodies at 4 Weeks after Last Dose of HZ/su Vaccine | 4 Weeks after Last Dose of HZ/su Vaccine (Week 12 for Vaccine, then Placebo Arm; Week 36 for Placebo, then Vaccine Arm)
  Antibody levels measured using patient blood samples.
Levels of Serum Varicella-Zoster Virus Anti-Glycoprotein E Antibodies at 24 Weeks after First Dose of HZ/su Vaccine | 24 Weeks after First Dose of HZ/su vaccine (Week 24 for Vaccine, then Placebo Arm; Week 48 for Placebo, then Vaccine Arm)
  Antibody levels measured using patient blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Saxena, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Amit Saxena (Amit.Saxena@nyulangone.org). The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Amit.Saxena@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.